CLINICAL TRIAL: NCT02854137
Title: Evaluation of the Irritation Potential of Sunscreen Products in Human Eyes
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Bayer (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Other
Other Study IDs: 18434
Record Dates: First submitted 2016-07-29; First posted 2016-08-03 (Estimated); Last update posted 2018-12-12 (Actual); Status verified 2018-12

CONDITIONS: Sunscreening Agents

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Sunscreen / Arm 1 (Experimental): Subjects will be escorted to a separate room for instillation of the test materials. Test materials will be instilled in immediate succession and with a randomized order of presentation. A trained technician will use the thumb and forefinger of one hand to retract the lower eyelid from the eyes of the subject forming sacs in the conjuntival tissue, apply one test product to one eye.
  Interventions: Drug: BAY987521
- Control (Other): A trained technician will use the thumb and forefinger of one hand to retract the lower eyelid from the other eyes of the subject forming sacs in the conjuntival tissue, apply control materials to this eye, follow the same procedure, using a new pipet tip or steriled dropper.
  Interventions: Drug: Control

INTERVENTIONS:
Drug: BAY987521 — 10 micro L of the appropriate test product is place into the lower conjunctival sac of the designated eye (Formulation code: Y49-103).
  Arms: Sunscreen / Arm 1
Drug: Control — 10 micro L of the appropriate controlled product is place into the lower conjunctival sac of the designated eye.
  Arms: Control

SUMMARY:
Evaluation of the human eye irritation potential of a test sunscreen formulation.

ELIGIBILITY:
Inclusion Criteria:

* Subjects must be healthy males or females between the ages of 18 to 60 years inclusive.
* Subjects do not wear contact lenses or willing to refrain from wearing them during the day of and day after the study.
* Subjects are willing to report any medications taken during the study and refrain from taking any medication during the study.
* Subjects are willing to have the test materials instilled into the eyes and follow all protocol requirements.

Exclusion Criteria:

* Subjects have ocular disease or peri-orbital dermatitis or trauma.
* Subjects have a systemic illness which contra-indicates participation.
* Subjects must not have a history of pre-existing sensitivity or other types of allergy to any eye products.
* Subjects must not have a history of allergies or sensitivities to cosmetics, toiletries, dermatological products, or any ingredients contained in the test or control products.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 23 (Actual)
Dates: Start 2015-10-14 (Actual); Primary Completion 2015-10-14 (Actual); Study Completion 2015-10-14 (Actual)

PRIMARY OUTCOMES:
Macroscopic evaluations for Lacrimation (score 0-4) | up to 1 hour post instillation
Macroscopic evaluations for Bulbar Conjuctiva Irritation (score 0-3) | up to 1 hour post instillation
Macroscopic evaluations of Palpebral Conjunctiva Irritation (score 0-3) | up to 1 hour post instillation
Subjective assessment of discomfort (score 0-4) | up to 1 hour post instillation

CONTACTS AND LOCATIONS:
Overall Officials: Bayer Study Director, Study Director — Bayer
Locations (1):
- St. Petersburg, Florida, United States